CLINICAL TRIAL: NCT07124559
Title: Phase I/II Dose Finding, Safety and Tolerability Study of Daily Rifapentine Combined With Isoniazid (1HP) for Tuberculosis Prevention in Children Less Than 13 Years of Age With and Without HIV
Brief Title: A Study of Daily Rifapentine Combined With Isoniazid (1HP) for Tuberculosis Prevention in Children Less Than 13 Years of Age With and Without HIV
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IMPAACT 2024; 38747 (Other: DAIDS Study ID)
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Tuberculosis
Keywords: HIV; Tuberculosis; Latent Tuberculosis
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — rifapentine; Isoniazid; dolutegravir

STUDY DESIGN:
Intervention Model Description: Cohort 1 will open to enrollment first and Cohort 2 will open following RPT dose confirmation in Cohort 1. Within each cohort, participants in all weight bands will be enrolled concurrently.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Children living without HIV (Experimental): Participants will be enrolled by weight bands across five weight groups.
  Interventions: Drug: Rifapentine; Drug: Isoniazid
- Cohort 2: Children living with HIV (Experimental): Participants will be enrolled by weight bands across five weight groups.
  Interventions: Drug: Rifapentine; Drug: Isoniazid; Drug: Dolutegravir

INTERVENTIONS:
Drug: Rifapentine — Dispersible Tablet administered orally
  Other Names: RPT
Drug: Isoniazid — Dispersible Tablet administered orally
  Other Names: INH
Drug: Dolutegravir — Tablets and Tablets for oral suspension administered orally
  Arms: Cohort 2: Children living with HIV

SUMMARY:
This study aims to find the proposed dose of Rifapentine (RPT) taken once daily with Isoniazid (INH) for 28 days to prevent tuberculosis (TB). The study will take place at multiple locations and children under 13 years old will be divided into two groups: one group will include children without HIV, and the other group will include children with HIV who are on antiretroviral treatment. Up to 144 children will participate, and participants in each group will be followed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A parent or legal guardian must be willing and able to give written permission for the child to participate in the study. If required by local policies, the child must also be willing and able to give written assent to participate. All sites must follow local policies and procedures.
2. Age requirements at entry:

   * Cohort 1: Children under 13 years old.
   * Cohort 2: Children aged 12 weeks to under 13 years old.
3. For Cohort 1 participants under 28 days old: The child must have been born at or after 37 weeks of pregnancy, as determined by the site investigator using parent/guardian report or medical records.
4. Weight requirements at entry:

   * Cohort 1: 3 kg to under 45 kg.
   * Cohort 2: 6 kg to under 45 kg.
5. HIV status:

   * Cohort 1: Must be living without HIV.
   * Cohort 2: Must be living with HIV.
6. At risk of TB disease, defined as meeting at least one of the following:

   * Having close contact with someone with infectious pulmonary TB within the past six months.
   * A positive tuberculin skin test (TST) or, for those over two years old, a positive interferon gamma release assay (IGRA) if TST is not available.
   * For Cohort 2 only: Living in a high TB burden area (≥ 60 TB cases per 100,000 people per year).
7. Normal or mild (grade 1 or 2) test results for the following at screening (within 21 days before entry):

   * ALT (liver enzyme)
   * Estimated glomerular filtration rate (kidney function)
   * Absolute neutrophil count (white blood cells)
   * Hemoglobin (red blood cells)
8. For Cohort 2 participants:

   * Must have been on antiretroviral therapy (ART) for at least 12 weeks before entry.
   * Must have been on a specific ART regimen (once-daily DTG and two NRTIs) for at least 14 days before entry.
   * Must have used the same formulation of DTG (tablet or dispersible tablet) for at least three days before entry.
   * Must agree to continue the same formulation of DTG for the study duration.
   * Must have an HIV-1 RNA level below 200 copies/mL at screening.
9. Must intend to stay in the same area for the study duration.
10. Must have access to at least one meal per day during the 28-day treatment period.

Exclusion Criteria:

1. The child has active TB, confirmed by medical records, parent/guardian report, or tests during screening, indicated by:

   * Currently being treated for active TB.
   * Symptoms like poor growth, poor weight gain, weight loss, cough for at least 11 days, or fever for at least eight days.
   * X-ray or CT scan showing TB.
   * Positive TB test results (e.g., culture, Xpert MTB/RIF Ultra, Truenat M.tb, other nucleic acid tests, urine tests).
2. The child has been exposed to an adult with drug-resistant TB (resistant to Rifampicin or Isoniazid) within the past six months.
3. The child has taken the following medications:

   * Daily Isoniazid in the 28 days before entry.
   * Any prohibited medications listed in the study within three days before entry.
4. The child has any of the following conditions:

   * Acute or chronic hepatitis.
   * Allergy to Isoniazid or rifamycins.
   * Porphyria.
   * Severe peripheral neuropathy.
5. The child has severe acute malnutrition (weight-for-height/length less than -3 z-scores of WHO standards). Note: Children who are stunted (height-for-age more than two standard deviations below WHO standards) are eligible.
6. For Cohort 2: The child has an active AIDS-defining opportunistic infection.
7. The child has started menstruation.
8. The child has taken NVP, EFV, lopinavir/ritonavir, and/or raltegravir within 14 days before entry.
9. The child has received long-term immunosuppressive therapy (more than eight days) within 30 days before entry. Note: Short courses of steroids (seven days or less) may be allowed with approval.
10. The child is a result of a multiple birth (e.g., twins, triplets).
11. The child has any other significant medical condition that would make participation unsafe, complicate data interpretation, or interfere with study objectives, as determined by the site investigator.

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Rifapentine (RPT) at specified time points among children with and without HIV | Through Day 28
Area Under the Curve (AUC)(0-inf) of RPT | Through Day 28
Maximum serum concentration (C(max)) of RPT | Through Day 28
Half-life (t1/2) of RPT | Through Day 28
Apparent oral clearance (CL/F) of RPT | Through Day 28
Apparent oral volume of distribution (V/F) of RPT | Through Day 28
Absorption rate (ka) of RPT | Through Day 28
Trough serum concentration (C(trough)) of DTG (Cohort 2 only) | At study entry, Day 28 and Day 42
CL/F of DTG (Cohort 2 only) | At study entry, Day 28 and Day 42
Proportion of participants experiencing Adverse Events (AEs) | Through Day 28
Proportion of participants experiencing Grade 3 or higher AEs | Through Day 28
Proportion of participants experiencing Grade 2 or higher AEs assessed as related to 1HP | Through Day 28
Proportion of participants experiencing Serious Adverse Events (SAEs) assessed as related to 1HP | Through Day 28
Proportion of participants experiencing AEs assessed as related to 1HP that led to permanent discontinuation of the regimen | Through Day 28

SECONDARY OUTCOMES:
Relative effects of significant covariates on RPT PK | Through Day 28
  Significant covariates include age, weight, sex, ethnicity, nutritional status, and HIV-1 status
Proportion of participants experiencing AEs | Through Day 168
Proportion of participants experiencing Grade 3 or higher AEs | Through Day 168
Proportion of participants experiencing Grade 2 or higher AEs assessed as related to 1HP | Through Day 168
Proportion of participants experiencing SAEs assessed as related to 1HP | Through Day 168
Participant and/or parent/guardian reported palatability and acceptability of 1HP regimen | At Day 1, Day 14, and Day 28
Number of occurrences of permanent discontinuation of 1HP regimen due to participant refusal to take 1HP or participant's parent/guardian decision to prematurely discontinue 1HP regimen | Through Day 168
Participant adherence to the 1HP regimen | Through Day 28
  Defined as having maintained at least 85% adherence to the 1HP regimen (24 doses) measured by observed and confirmed dosing and participant/parent/guardian report.
Proportion of participants experiencing Grade 2 or higher AEs assessed as related to DTG (Cohort 2 only) | Through Day 42
Proportion of participants experiencing SAEs assessed as related to DTG (Cohort 2 only) | Through Day 42
Proportion of participants experiencing AEs assessed as related to DTG that led to permanent discontinuation of the regimen (Cohort 2 only) | Through Day 42
Number of participants with HIV-1 RNA less than 200 copies/mL (Cohort 2 only) | At Day 42

CONTACTS AND LOCATIONS:
Locations (11):
- Botswana (2):
  - Gaborone (Site ID: 12701), Gaborone
  - Molepolole (Site ID: 12702), Gaborone
- Les Centres GHESKIO (Site ID: 30022), Port-au-Prince, Haiti
- Kenya Medical Research Institute, Walter Reed Project Clinical Research Center (Site ID: 5121), Kericho, Kenya
- Thailand (2):
  - Siriraj Hospital, Mahidol University (Site ID: 5115), Bangkok, Bangkoknoi
  - Chiangrai Prachanukroh Hospital (Site ID: 5116), Chiang Rai
- Uganda (2):
  - Baylor-Uganda (Site ID: 31798), Kampala
  - MU-JHU Care Limited (Site ID: 5126), Kampala
- Zimbabwe (3):
  - Harare Family Care (Site ID: 31890), Belgravia, Harare
  - Seke North (Site ID: 30306), Belgravia, Harare
  - St Mary's (Site ID: 30303), Chitungwiza

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data